CLINICAL TRIAL: NCT05012917
Title: A Randomized Controlled Trial a Dyad Approach to Symptom Screening (Co-SSPedi) vs. Proxy-report (Proxy-SSPedi) and Self-report (SSPedi or Mini-SSPedi) for Pediatric Patients Receiving Cancer Treatments
Brief Title: Parent/Child Dyad Approach to Symptom Screening for Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000076793
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Pediatric Cancer; Quality of Life; Symptom Screening
Keywords: Pediatric Oncology; Randomized Controlled Trial; Symptom Screening; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized cross-over study that involves a single interview where the primary analysis will involve the first period only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient/Proxy-SSPedi Administered First (Other): Parent/child dyads will complete self-report SSPedi/mini-SSPedi and proxy-SSPedi as the first "period" and then co-SSPedi as a second "period".
  Interventions: Other: Patient/Proxy-SSPedi; Other: Co-SSPedi
- Co-SSPedi Administered First (Other): Parent/child dyads will complete co-SSPedi as the first "period" and then self-report SSPedi/mini-SSPedi and proxy-SSPedi as a second "period".
  Interventions: Other: Patient/Proxy-SSPedi; Other: Co-SSPedi

INTERVENTIONS:
Other: Patient/Proxy-SSPedi — SSPedi and Mini-SSPedi: SSPedi is a symptom assessment scale for children 8-18 years of age that includes 15 symptoms considered most important by children receiving cancer treatment or HSCT, their parents and healthcare professionals. Each symptom is rated on a 5-point Likert scale consisting of 0="not at all bothered", 1="a little", 2="medium", 3="a lot" and 4="extremely bothered". The recall period is yesterday or today.
  Mini-SSPedi was developed for children 4-7 years of age and is comprised of the same 15 symptoms. Mini-SSPedi has a recall period of today with a 3-point Likert scale consisting of 0="not at all bothered", 2="medium" and 4="extremely bothered'. So, the anchors and mid-point are identical to SSPedi. A faces-type scale accompanies the response options and the symptom descriptions are simplified.
  Proxy-SSPedi: Proxy-SSPedi is identical to SSPedi except that the leading question refers to "your child" rather than "you". It is designed for children 2-18 years of age.
Other: Co-SSPedi — Co-SSPedi: Co-SSPedi is based upon either SSPedi (age 8-18) or mini-SSPedi (age 4-7).
  Co-SSPedi is meant to be completed by both child and parent together. The format and wording is identical to self-report SSPedi and mini-SSPedi (depending on child age) to maximize the ability of the child to participate in symptom reporting.
  The approach uses written instruction that asks the dyad who will hold the device and enter the agreed-upon scores. The instruction then asks one member to read the leading question, each symptom and response options out loud. The child answers how bothered they are by that symptom out loud. The parent then states if they agree or they can offer a different answer. If the answer is different, the instruction asks the dyad to discuss until they agree upon an answer. The agreed-upon answer is then entered into co-SSPedi. This process is repeated for the remaining 14 symptoms.

SUMMARY:
Symptoms are common and often severely bothersome in pediatric patients receiving cancer treatments. In order to measure the extent of bothersome symptoms, the Symptom Screening in Pediatrics Tool (SSPedi) was developed. It is reliable, valid and responsive to change in pediatric patients aged 8-18 years receiving cancer treatments. Mini-SSPedi was developed for children 4-7 years and exhibits face and content validity. These instruments were developed to address the lack of appropriate symptom screening tools for this population. They are available in both self-report and proxy-report formats.

Differences between child self-report and parent proxy-report quality of life (QoL) scores have been well described in pediatric populations. There has been increasing recognition that each reporter may have unique and valid perspectives. This has led to a suggestion to collect both child and parent report when possible.

When used in clinical care, obtaining both child and parent report will commonly not be feasible. There are settings in which children will not be willing to independently report symptoms, such as when they are very ill. Unfortunately, it is particularly in this setting that obtaining symptoms reports is crucial. While young children may be able to independently report symptoms on a single occasion in the context of a carefully conducted research study, they are less likely to be able to repeatedly and independently report their symptoms. Finally, the burden and logistical complexity of separate child and parent reporting would be associated with considerable challenges for clinical implementation.

In considering how routine symptom screening could be implemented into clinical practice, we hypothesized that a dyad approach, where SSPedi is completed by both the child and parent together, may be one way to address these challenges. Consequently, we developed and finalized the approach to co-SSPedi administration, with instruction that is easy to understand, resulting in dyads completing co-SSPedi correctly.

To understand the relationships between the available forms of SSPedi (co-SSPedi, proxy-SSPedi and SSPedi), outstanding questions are how co-SSPedi scores compare to either proxy-report or self-report SSPedi and whether the co-SSPedi administration approach increases or decreases score variability. This study is designed to address these questions.

DETAILED DESCRIPTION:
The overall goal of this randomized, cross-over study is to describe the distribution of co-SSPedi scores when compared to proxy-report and self-report SSPedi or mini-SSPedi scores. We hypothesize co-SSPedi would be significantly different than proxy-report and self-report SSPedi with respect to score distribution, and would have decreased symptom score variability.

Aim 1: To compare the mean co-SSPedi scores vs. proxy-SSPedi for pediatric patients with cancer or HSCT recipients who are 4-18 years of age.

Aim 2: To compare the mean co-SSPedi scores vs. self-report SSPedi/mini-SSPedi scores for pediatric patients with cancer or HSCT recipients who are 4-18 years of age.

Aim 3: To describe differences in interquartile range, standard deviation and range between co-SSPedi scores vs. proxy-report or self-report SSPedi/mini-SSPedi scores.

Aim 4: To obtain qualitative feedback about the experience of completing symptom screening together vs. separately from pediatric patients and their parents

Overall Strategy

This study is a randomized cross-over study that involves a single interview where the primary analysis will involve the first period only. This study will be conducted at a single center, The Hospital for Sick Children (SickKids) in Toronto. The study population will comprise participants across all oncology and HSCT sections within the Division of Haematology/Oncology.

Research Methods

Eligibility: This study will enroll child-parent dyads. We will include English-speaking dyads of a child and a guardian, where the child is between 4-18 years of age and has a diagnosis of cancer or is a hematopoietic stem cell transplant (HSCT) recipient. Exclusion criteria will be illness severity, cognitive disability or other impairment that precludes completion of co-SSPedi, SSPedi/mini-SSPedi or proxy SSPedi according to the primary healthcare team. Both inpatients and outpatients will be eligible.

Procedures: The instruments will be administered on an electronic platform. Each dyad will complete both co-SSPedi as one "period" and then self-report SSPedi/mini-SSPedi and proxy-SSPedi as a second "period". Both "periods" will occur during the same dyad encounter. The order of periods will be randomized, resulting in two groups based upon the approach used in the first period. The allocation sequence will be computer generated and will be concealed from all participants, healthcare providers and research team members. Consenting participants will be randomized 1:1 to co-SSPedi administration first vs. self-report/proxy-report first using permuted block sizes and stratified by relapse status (yes vs. no), age (4-7, 8-10, 11-14 and 15-18 years) and outpatient/ inpatient at time of interview as our previous data suggested that these factors were the most strongly associated with higher total SSPedi scores.

The dyad will complete the randomized approach first and then will proceed to the alternate approach. After the second period, qualitative feedback will be elicited using a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Child and guardian both understand English
* Child is 4 to 18 years of age
* Child has diagnosis of cancer or is a hematopoietic stem cell transplant (HSCT) recipient
* Child is inpatient or outpatient

Exclusion Criteria:

* Participants who have illness severity,
* cognitive disability, or
* visual impairment that preclude utilization of co-SSPedi, SSPedi/mini-SSPedi or proxy SSPedi according to the primary healthcare team

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 420 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Symptom Screening in Pediatrics Tool (SSPedi) total score | Immediately after the intervention
  The total SSPedi score is a measure that reflects the total burden of bothersome symptoms experienced.
  Total unweighted scores will be calculated for co-SSPedi, SSPedi/mini-SSPedi and proxy-SSPedi. The scoring for all instruments is identical. Each item's Likert score ranges from 0 (no bother) to 4 (worst bother); Likert scores are summed for a total score that ranges from 0 (none) to 60 (worst possible).

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dupuis LL, Johnston DL, Baggott C, Hyslop S, Tomlinson D, Gibson P, Orsey A, Dix D, Price V, Vanan M, Portwine C, Kuczynski S, Spiegler B, Tomlinson GA, Sung L. Validation of the Symptom Screening in Pediatrics Tool in Children Receiving Cancer Treatments. J Natl Cancer Inst. 2018 Jun 1;110(6):661-668. doi: 10.1093/jnci/djx250. PMID 29272441
- [Background] Hyslop S, Dupuis LL, Baggott C, Dix D, Gibson P, Kuczynski S, Johnston DL, Orsey A, Portwine C, Price V, Spiegler B, Tomlinson D, Vanan M, Tomlinson GA, Sung L. Validation of the Proxy Version of Symptom Screening in Pediatrics Tool in Children Receiving Cancer Treatments. J Pain Symptom Manage. 2018 Jul;56(1):107-112. doi: 10.1016/j.jpainsymman.2018.03.025. Epub 2018 Apr 6. PMID 29630923